CLINICAL TRIAL: NCT03653286
Title: Effect of Physical Training With Neuromuscular Eletroestimulation in Torque and Performance of Long Distance Recreational Runners Randomized Clinical Trial
Brief Title: Neuromuscular Eletroestimulation in Torque for Long Distance Recreational Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Richard Eloin Liebano, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNICIDAGRREM14
Record Dates: First submitted 2018-08-26; First posted 2018-08-31 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Torque
Keywords: Neuromuscular Eletrical Stimulation; Torque; Runners
MeSH Terms: interventions — Jogging

STUDY DESIGN:
Intervention Model Description: The runners will be randomized into two groups, being: control group (CG) - will perform only run and intervention group (GI) - using the medium-frequency alternating current and run.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigations of the peak muscle torque, analysis of ventilatory anaerobic thresholds, running economy and maximal oxygen consumption will be performed by a blind investigator. Data analysis will be performed by a blind investigator in the control and intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES and Run (Experimental): NMES and run
  Interventions: Other: NMES and Run
- Only Run (Other): Only Run
  Interventions: Other: Only Run

INTERVENTIONS:
Other: NMES and Run — NMESIn this exercise protocol for quadriceps strengthening using NMES, the medium-frequency alternating current (1KHz with 10% of the work cycle) 4 will be used. The total daily training time is 900sec (15min), it is expected to perform 45 contractions per training, with three workouts per week for six weeks.
  RUN: It will be allowed to carry out training drills that comprise 15-40Km per week, being allowed a minimum of 2 and a maximum of 3 training sessions per week, not being able to carry out drills of explosion and during each training must be covered at least 5km and at most 15km. These limitations were based on the American College of Sports Medicine (ACSM) cardiorespiratory training guidelines to minimize confounders of cardiopulmonary performance.
  Arms: NMES and Run
Other: Only Run — RUN: It will be allowed to carry out training drills that comprise 15-40Km per week, being allowed a minimum of 2 and a maximum of 3 training sessions per week, not being able to carry out drills of explosion and during each training must be covered at least 5km and at most 15km. These limitations were based on the American College of Sports Medicine (ACSM) cardiorespiratory training guidelines to minimize confounders of cardiopulmonary performance.
  Arms: Only Run

SUMMARY:
Introduction: The use of neuromuscular electrical stimulation (NMES) in athlete training has become an increasingly common feature among competition teams. Among the main benefits of NMES are the increase in muscular strength and improvement in athletes' performance. Surveys demonstrate the benefits of basketball, volleyball, soccer, swimmers and Olympic lifters using NMES, but no studies have been conducted on runners. Objectives: To evaluate the effects of 6 weeks of training with NMES, on knee peak torque (PT), ventilatory anaerobic threshold, maximum oxygen consumption (VO2max) and running economy in recreational runners. Methods: Randomized clinical trial involving 30 long distance runners, being randomly distributed in 2 groups of 15 participants each. All individuals will perform isokinetic evaluation of the lower limbs and ergospirometry. After these evaluations, all athletes will perform the same running training (CT), in addition to the CT the intervention group will perform NMES on the knee extensors 3 times a week for 15 minutes.

DETAILED DESCRIPTION:
Participants who meet the eligibility criteria will be invited to participate in the study and, after signing the informed consent form, will perform initial clinical evaluation and will be randomized into two groups, being: control group (CG) and intervention group (GI) - using the medium-frequency alternating current. Each group will consist of 15 subjects who will have as dependent variables, the evaluation of the following items: peak muscle torque, analysis of ventilatory anaerobic thresholds, running economy and maximal oxygen consumption.

The intervention with the NMES will be considered as an independent variable. All groups will have the dependent variables evaluated before and after the intervention, which will consist of 18 sessions (6 weeks). The NMES training will be performed 3 times a week and will never be applied for two consecutive days, as shown in the flowchart All individuals, being they of the CG or the GI will perform a running training (TC), between 15 and 40 km per week and will be guided how to perform them, and the GI patients will perform a muscle strengthening protocol with NMES, which will be carried out in a specific place and prepared for intervention, in addition to the TC.

ELIGIBILITY:
Inclusion Criteria:

* Included will be male individuals, aged 30 to 45 years
* recreational funders, who have been performing the activity for at least 1 year.
* Totaling at least 15km and a maximum of 40km of training per week,
* Who do not use NMES for the purpose of muscle training.

Exclusion Criteria:

* Subjects who present muscle injuries and / or joint injuries in the lower limbs (LMI) in the last 6 months can't be part of the study.
* Who are unable to perform the isokinetic test
* Who are unable to do ergospirometric test,
* Who meet the contraindications criteria of NMES

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Included will be male individuals, aged 30 to 45 years, recreational runners, who have been performing the activity for at least 1 year, totaling at least 15km and a maximum of 40km of training per week, who do not use NMES for the purpose of muscle training.
  Subjects who suffer muscle injuries and / or joint injuries in the lower limbs (LMW) during the 6 weeks of training, Subjects who present muscle injuries and / or joint injuries in the lower limbs (LMI) in the last 6 months can't be part of the study.
Enrollment: 30 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Isokinetic dynamometer | 6 weeks
  The computerized isokinetic muscle evaluation will be performed in the Cybex Norm isokinetic dynamometer (Cybex International, Inc., Ronkonkoma, LI, New York), at the Physiotherapy Clinic of Universidade Cidade de São Paulo (UNICID). The movement performed during the test will be that of isometric, concentric and eccentric extension of the two knees, to measure peak torque, using angulations of 90 to 60 degrees of knee and 3 maximum voluntary contractions.

SECONDARY OUTCOMES:
Maximum oxygen consumption | 6 weeks
  Prior to the test, subjects will lie down for 10 minutes for initial ventilatory data and heart rate (HR) records. The test protocol will consist of running on a treadmill (ATL Model, Inbrasport Ltda, Brazil), with an initial velocity of 6km / h, followed by increments of 1km / h every 1min until voluntary exhaustion of the subjects.
  Ventilatory parameters will be collected during rest and continuously throughout the tests, at each respiratory cycle, and analyzed in averages of 20sec through a computerized gas analyzer (model VO2000; Inbrasport Ltda, Brazil). The gas analyzer shall be calibrated to the volume and standard concentration of gases immediately before the first test of the day and re-calibrated after each test as per manufacturer's standardization.
Racing economy | 6 weeks
  The running economy on a horizontal treadmill will be measured in 3 speeds in the order indicated: 2.68, 3.13 and 3.58 m · s-1 (9.6, 11.3 and 12.9 km · h-1, respectively). The guy will run for 6 minutes at each speed and rest between runs. The VO2 per minute will be measured during each of the last 3 minutes of each race. The mean of the difference of the 2 values will be used as a measure of the running economy.
  The economy will be expressed in meters per milliliter of oxygen consumed per kilogram of body weight (m / ml-1 / kg-1). This unit allows comparisons at various running speeds, and has a conceptual advantage in that the numerical values are directly related to the economy (ie, the higher the number the better the economy).
Analysis of Ventilatory Anaerobic Threshold | 6 weeks
  The LAVs will be determined from ventilatory equivalents (VE / VO2 and VE / VCO2), final expired fractions (FEO2 and FECO2) and respiratory quotient (QR), and expressed as VO2 (in ml / kg / min). The LAV1 will correspond to the lowest value of EV / VO2 before its continuous increase associated with the beginning of the abrupt and continuous increase of the QR.
  The LAV2 will correspond to the point at which the nonlinear increases of VE / VO2, VE / VCO2 and FEO2 will coincide with the decrease of FECO2. Immediately after the 18th training session, the patients will be re-evaluated and submitted to all the procedures described for isokinetic evaluation and ergospirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, Study Director — Universidade Cidade de Sao Paulo
Locations (1):
- UNICID, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No